CLINICAL TRIAL: NCT02143661
Title: eValuatIon of The ALl New Environment for crITicallY Ill Patients (VITALITY)
Status: Completed | Type: Observational
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow - Klinikum, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: Vitality
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Intensive Care Unit Environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critically ill patients in the newly designed ICU rooms: Critically ill patients treated in one of the newly designed ICU rooms.
- Critically ill patients in the conventional ICU rooms: Critically ill patients treated in one of the conventional rooms on the same ICU.

SUMMARY:
The purpose of this prospective observational study is to investigate if mechanically ventilated patients who are treated in one of the new intensive care unit (ICU) rooms have less delirium compared to patients who are treated in the conventional rooms on the same ICU. The investigators will further evaluate the impact on sleep quality, circadian rhythm, global cognitive function and general outcome parameters.

The investigators recorded light and noise conditions in the ICU rooms before start of the redesigning process (subproject light and noise in the intensive care unit (LiNo-ICU)). The investigators will compare data regarding light and noise in the ICU rooms before and after the redesigning process (non-patient related data; ethical vote amendment 08.05.2014).

DETAILED DESCRIPTION:
Delirium is one of the most frequently seen brain organ dysfunctions in the intensive care unit (ICU). Depending on the ICU population, up to 87% have delirium at some point during their critical illness. Patients with delirium have a 3fold increased risk of dying compared to patients without delirium. Studies could show that sedation is the most common independent risk factor for transitioning to delirium. However, the no-sedation approach is often challenging. ICU patients who are not sedated often develop severe anxiety and agitation. These symptoms are often treated with sedatives that have delirogenic side effects.

One of the major reasons for anxiety and agitation of patients is the ICU environment which causes distress. The feelings of being surveyed all the time by monitors, being exposed to different kinds of machinery or equipment which sometimes do not work properly are major stressors.

The objective of the interdisciplinary research project "Parametrische (T)Raumgestaltung" was the development of two redesigned intensive care rooms that help to reduce patients' anxiety, helplessness and stress through a holistic architectural approach. The patient's perception and needs, his or her obvious feelings of helplessness and fear are the starting point for a concept that is able to reduce stress factors such as functional and purely technical environment, insufficient lighting conditions and noise. Minimizing or eliminating these common stress factors in the ICU could reduce the need for sedatives and thereby reducing the incidence of ICU delirium.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age ≥ 18 years
* Expected intensive Care unit stay ≥ 48 hours
* Invasive mechanical ventilation or non-invasive mechanical ventilation (with positive ventilation pressure >6 hours/day and high flow >30 liters) on the day of intensive care unit admission

Exclusion Criteria:

* Participation in other clinical studies 10 days before study inclusion and during the study period
* Patients with psychiatric diseases
* Patients with a history of stroke and known residual cognitive deficits
* Patients with a history of cardiopulmonary arrest or pulseless electric activity with cardiopulmonary resuscitation followed by therapeutic hypothermia during entire hospital stay
* Analphabetism
* Anacusis or Hypoacusis with hearing aid device, Amaurosis
* Non-German speaking
* Allergies to any substance of the electrode fixing material
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* History of sleep disorders
* History or suspicion of hypoxic brain damage (e.g. intracranial bleeding)
* History or suspicion of elevated intracranial pressure in the last 7 days before study inclusion
* Patients with an open chest after cardiac surgery
* The informed consent of the patient or the subject's legally acceptable representative can´t be obtained in time
* Patient has a power of attorney or patient's provision, where he/she refuses participation in any clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of intensive care unit delirium | Participants will be followed up to 10 days after intensive care unit admission
  Delirium will be measured with the Confusion Assessment Method for the intensive care unit (CAM-ICU)

SECONDARY OUTCOMES:
Circadian plasma melatonin level | Participants will be followed up to 10 days after intensive care unit admission
  Plasma melatonin levels will be assessed in a maximum of three 24-hour periods. Blood samples will be collected every 4 hours within each series of measurements.
Circadian plasma cortisone level | Participants will be followed up to 10 days after intensive care unit admission
  Plasma cortison levels will be assessed in a maximum of three 24-hour periods. Blood samples will be collected every 4 hours within each series of measurements.
Gene expression of clock genes in blood monocytes | Participants will be followed up to 10 days after intensive care unit admission
  Clock gene levels in blood monocytes will be assessed in a maximum of three 24-hour periods. Blood samples will be collected every 4 hours within each series of measurements.
Cholinesterase activity in blood | Participants will be followed up to 10 days after intensive care unit admission
  The Activity of Cholinesterase will be measured at least once a day, maximum three times a day.
Core body temperature | Participants will be followed up to 10 days after intensive care unit admission
  Temperature will be measured continuously during those days
Severity of intensive care unit delirium | Participants will be followed up to 10 days after intensive care unit admission
  Severity of delirium will be measured with the Intensive Care Delirium Screening Checklist (ICDSC)
Severity of anxiety | Participants will be followed up to 10 days after intensive care unit admission
  Severity of anxiety will be measured with the Faces Anxiety Scale (FAS)
Post-Traumatic Stress Disorder (PTSD) | Up to 3 and 6 months after intensive care unit discharge
  At intensive care unit discharge, at hospital discharge, 3 and 6 months after intensive care unit discharge Post-Traumatic Stress Disorder Incidence will be measured with the PTSS-14 Scale
Barthel Index | Up to 3 and 6 months after intensive care unit discharge
  Barthel Index will be measured at hospital discharge, 3 and 6 months after intensive care unit discharge.
Health Related Quality of Life | Up to 3 and 6 months after intensive care unit discharge
  At 3 and 6 months after intensive care unit discharge. Health Related Quality of Life will be measured with the Short Form questionnaire (SF-36)
Global cognition and executive function | Up to 3 and 6 months after intensive care unit discharge
  At intensive care unit discharge, at hospital discharge, 3 and 6 months after intensive care unit discharge.
Polysomnography | Participants will be followed up to 10 days after intensive care unit admission
  Polysomnography will be performed for a maximum of three 24-hour periods. Polysomnography will start after the 1st, 3rd and 5th night of intensive care unit admission.
Subjective sleep quality | Participants will be followed up to 10 days after intensive care unit admission
  Subjective sleep quality will be assessed with the Sleep Questionnaire SF-A from Collegium Internationale Psychiatriae Scalarum at morning of 2nd, 4th and 6th day of study participation.
Duration of mechanical and non-mechanical ventilation | Participants will be followed for the duration of intensive care stay, an expected average of 1 week
Intensive care unit length of stay | Participants will be followed for the duration of intensive care stay, an expected average of 1 week
Hospital length of stay | Participants will be followed for the duration of hospital length of stay, an expected average of 3 weeks
Level of sedation | Participants will be followed up to 10 days after intensive care unit admission
  Level of sedation will be measured with the Richmond Agitation-Sedation-Scale (RASS)
Sedation goal adherence | Participants will be followed up to 10 days after intensive care unit admission
  Adherence of optimal sedation level measured by Richmond Agitation-Sedation-Scale (RASS)
Pain level | Participants will be followed up to 10 days after intensive care unit admission
  Pain level will be measured with the Numeric Rating Scale (NRS), or the Visualized Numeric Rating Scale (NRS-V) or the Faces Pain Scale-Revised (FPS-R) or the Behavioral Pain Scale (BPS) or the Behavioral Pain Scale for Non- Intubated (BPS-NI).
Amount of administered opioids | Participants will be followed up to 10 days after intensive care unit admission
Amount of administered benzodiazepines | Participants will be followed up to 10 days after intensive care unit admission
Amount of administered antipsychotics | Participants will be followed up to 10 days after intensive care unit admission
Sepsis/Septic shock | Participants will be followed up to 10 days after intensive care unit admission
Sequential Organ Failure Assessment (SOFA-Score) | Participants will be followed up to 10 days after intensive care unit admission
Simplified Acute Physiology Score (SAPS II) | Participants will be followed up to 10 days after intensive care unit admission
Therapeutic Intervention Scoring System (TISS-28) | Participants will be followed up to 10 days after intensive care unit admission
Acute Physiological and Chronic Health Evaluation (APACHE II) | Participants will be followed up to 10 days after intensive care unit admission
Sleep-wake-behavior monitoring | Participants will be followed up to 10 days after intensive care unit admission
  Sleep-wake-behavior using actigraphy will be assessed continuously.
Light levels | Participants will be followed up to 10 days after intensive care unit admission
  Light levels will be measured continuously.
Light frequencies | Participants will be followed up to 10 days after intensive care unit admission
  Light frequencies will be measured continuously.
Noise levels | Participants will be followed for 10 days after intensive care admission
  Noise levels will be measured continuously.
Patients´ perception of the room and light environment | Participants will be followed for 10 days after intensive care admission
Hospital mortality | Up to 6 months
Multiplex-Genexpression analysis | Participants will be followed up to 10 days after intensive care unit admission
  Ncounter neuroinflammation and micro rna panel are analysed

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charité University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow - Klinikum, Charité- Universitätsmedizin, Berlin, Germany

REFERENCES:
- [Derived] Schmidt S, Heinrich M, Wernecke KD, Spies C, Hancke L, Mueller A, Luetz A. Modification in ICU design may influence circadian serum cholinesterase activities: a proof-of-concept pilot study. Intensive Care Med Exp. 2024 Dec 23;12(1):120. doi: 10.1186/s40635-024-00709-5. PMID 39715945
- [Derived] Spies C, Piazena H, Deja M, Wernecke KD, Willemeit T, Luetz A; ICU Design Working Group. Modification in ICU Design May Affect Delirium and Circadian Melatonin: A Proof of Concept Pilot Study. Crit Care Med. 2024 Apr 1;52(4):e182-e192. doi: 10.1097/CCM.0000000000006152. Epub 2023 Dec 19. PMID 38112493